CLINICAL TRIAL: NCT02627287
Title: A Comparative Trial Focusing on Injections With the Medical Device DV3316 Pen-injector Versus FlexPen
Brief Title: A Comparative Trial Focusing on Injections With the Medical Device DV3316 Pen-injector Versus FlexPen®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: INS-4208; 2014-004802-13 (EudraCT Number); U1111-1163-5039 (Other: WHO)
Record Dates: First submitted 2015-11-27; First posted 2015-12-10 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DV3316 pen-injector (Experimental)
  Interventions: Device: DV3316 pen-injector; Drug: placebo
- FlexPen® (Active Comparator)
  Interventions: Device: FlexPen®; Drug: placebo

INTERVENTIONS:
Device: FlexPen® — For subcutaneously (s.c. under the skin) injection.
  Arms: FlexPen®
Device: DV3316 pen-injector — For subcutaneously (s.c. under the skin) injection.
  Arms: DV3316 pen-injector
Drug: placebo — For subcutaneously (s.c. under the skin) injection

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare Injections with the Medical Device DV3316 Pen-injector versus FlexPen®.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-74 years (both included) at the time of signing informed consent
* T1DM (Type 1 Diabetes Mellitus) or T2DM (Type 2 Diabetes Mellitus) (as diagnosed clinically) at least 12 months prior to screening
* Daily self-injection(s) with anti-diabetic drug (insulin or Glucagon-Like Peptide-1 (GLP- 1) analogues) in pen-injector or vial/syringe for at least 12 months
* Caucasians
* Body Mass Index (BMI) at least 18.5 kg/m^2

Exclusion Criteria:

* Known or suspected hypersensitivity to test placebo solution incl. m-cresol and phenol or related products (placebo)
* Female who is pregnant,, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice)
* Known urticaria factitive or abnormal reactions to mechanical trauma
* Haemophilia and any diseases affecting blood coagulation
* Anti-coagulant or inhibitors of platelet aggregation treatment on the day of the visit
* Intake of any pain-relieving or analgesic drugs on the day of the site visit
* Skin diseases and infections of the skin in the injection site areas (abdomen and thighs)
* Lipodystrophia in the injection site areas (abdomen and thighs)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2016-02-25 (Actual)

PRIMARY OUTCOMES:
Injection success (full dose delivered s.c.) (yes/no) | By assessment that the dose counter has returned to "0" (EoD confirmation) for the DV3316 pen-injector and for FlexPen® at least 6 seconds after the dose counter has returned to "0"

SECONDARY OUTCOMES:
Subjects' confidence in injection completion (delivery of correct, full dose) | Injection completed within 2 minutes after needle insertion
Amount of liquid on the skin (placebo solution or tissue fluid) | Injection completed within 2 minutes after needle insertion
Subjects' reaction time | Injection completed within 2 minutes after needle insertion
Subjects evaluation of pen-injector experience | Injections completed within 2 minutes of needle insertion
Number of technical complaints | Day 1
Number of adverse device effects | Day 1
Grading of bleeding, redness, bruising and swelling at the site of injection | Within 10 minutes after completion of injection
Grading of bleeding, redness, bruising and swelling at the site of injection | 1 hour after completion of injection

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Germany (2):
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Neuss

REFERENCES:
- [Result] Tang H, Li G, Zhao Y, Wang F, Gower EW, Shi L, Wang T. Comparisons of diabetic retinopathy events associated with glucose-lowering drugs in patients with type 2 diabetes mellitus: A network meta-analysis. Diabetes Obes Metab. 2018 May;20(5):1262-1279. doi: 10.1111/dom.13232. Epub 2018 Feb 23. PMID 29369494
- [Result] Zijlstra E, Coester HV, Heise T, Plum-Morschel L, Rasmussen O, Rikte T, Pedersen LK, Qvist M, Sparre T. Injecting without pressing a button: An exploratory study of a shield-triggered injection mechanism. Diabetes Obes Metab. 2018 May;20(5):1140-1147. doi: 10.1111/dom.13203. Epub 2018 Jan 25. PMID 29369493
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com